CLINICAL TRIAL: NCT00003304
Title: Second Line Chemotherapy With Temozolomide in Recurrent Oligodendroglial Tumors After PCV-Chemotherapy
Brief Title: Temozolomide in Treating Patients With Recurrent Oligodendroglial Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-26972; EORTC-26972
Record Dates: First submitted 1999-11-01; First posted 2004-08-26 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult oligodendroglioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma | interventions — Temozolomide

INTERVENTIONS:
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of temozolomide in treating patients with recurrent oligodendroglial tumors following combination chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and duration of response in oligodendroglial tumors to temozolomide treatment in patients with progressive disease during or after procarbazine/lomustine/vincristine (PCV) chemotherapy. II. Determine the feasibility and toxicity of temozolomide chemotherapy following PVC chemotherapy in these patients.

OUTLINE: This is an open label, multicenter trial. Temozolomide is administered orally on days 1-5 of each 4-week course; treatment continues for a maximum of 12 courses. Patients are followed every 2 months for the first 6 months and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 16-29 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven oligodendroglioma or oligoastrocytoma (with at least 25% oligodendroglial elements) Recurrent or progressive disease following both radiotherapy and procarbazine/lomustine/vincristine chemotherapy (or other nitrosoureas-based chemotherapy) Contrast enhancing, measurable disease (at least one lesion measuring at least 1 cm) by CT or MRI required Within 2 weeks prior to study treatment Within 3 days following concurrent surgery for the recurrence Steroid doses stable or decreasing for at least 2 weeks prior to scan No extracranial disease

PATIENT CHARACTERISTICS: Age: 18-69 Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.25 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2 times ULN AST/ALT no greater than 2 times ULN Renal: Creatinine no greater than 1.25 times ULN Creatinine clearance at least 60 mL/min Other: Not pregnant or lactating Effective contraception required of fertile women No diseases interfering with follow-up

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No more than one prior chemotherapy regimen At least 4 weeks since prior chemotherapy Prior nitrosourea required At least 6 weeks since nitrosourea Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics More than 3 months since radiotherapy Surgery: Not specified Other: No concurrent treatment with other investigational agents or other antitumor agents

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 1998-04; Primary Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. van Den Bent, MD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (37):
- Kaiser Franz Josef Hospital, Vienna (Wien), Austria
- Hopital Universitaire Erasme, Brussels, Belgium
- Rigshospitalet, Copenhagen, Denmark
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Turku University Central Hospital, Turku
- France (13):
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier Universitaire de Bicetre, Le Kremlin-Bicêtre
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
  - CHU de Nancy - Hopital Neurologique, Nancy
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Hopital Pasteur, Nice
  - Centre Antoine Lacassagne, Nice
  - C.H.R. de Nimes - Hopital Caremeau, Nîmes
  - CHU Pitie-Salpetriere, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Universitaetsklinikum Benjamin Franklin, Berlin
  - Neurologische Klinik der Henriettenstiftung, Hanover
  - Universitaetsklinikum Tuebingen, Tübingen
- National Institute of Neurosurgery, Budapest, Hungary
- Italy (2):
  - Azienda Ospedaliera di Padova, Padova (Padua)
  - Universita Degli Studi di Torino, Torino
- Netherlands (9):
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - St. Radboud University Hospital, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
  - St. Elisabeth Ziekenhuis, Tilburg
  - Dr. Bernard Verbeeten Instituut, Tilburg
  - Academisch Ziekenhuis Utrecht, Utrecht
- Instituto Portugues de Oncologia de Francisco Gentil, Lisbon, Portugal
- Umea Universitet, Umeå, Sweden
- United Kingdom (2):
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland

REFERENCES:
- [Background] Kouwenhoven MC, Kros JM, French PJ, Biemond-ter Stege EM, Graveland WJ, Taphoorn MJ, Brandes AA, van den Bent MJ. 1p/19q loss within oligodendroglioma is predictive for response to first line temozolomide but not to salvage treatment. Eur J Cancer. 2006 Oct;42(15):2499-503. doi: 10.1016/j.ejca.2006.05.021. Epub 2006 Aug 17. PMID 16914310
- [Result] van den Bent MJ, Chinot O, Boogerd W, Bravo Marques J, Taphoorn MJ, Kros JM, van der Rijt CC, Vecht CJ, De Beule N, Baron B. Second-line chemotherapy with temozolomide in recurrent oligodendroglioma after PCV (procarbazine, lomustine and vincristine) chemotherapy: EORTC Brain Tumor Group phase II study 26972. Ann Oncol. 2003 Apr;14(4):599-602. doi: 10.1093/annonc/mdg157. PMID 12649108